CLINICAL TRIAL: NCT07303439
Title: Randomised Trial of Dual Device Treatment Involving Drug-coated Balloon Angioplasty and Drug-eluting Stent Implantation Compared to Single Device Treatments in Patients With Diabetes Mellitus
Acronym: DUBSTENT-DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Cardiovascular Research Institute Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 25183A001
Record Dates: First submitted 2025-06-13; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Coronary Arterial Disease (CAD); de Novo Coronary Lesions; De Novo Stenosis
Keywords: Diabetes Mellitus; Coronary Artery Disease; Drug-coated Balloon; Drug-Eluting Stent; Target Vessel Failure
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Patient's will be randomised to one of three arms, which include:
  1. . Drug-coated balloon in combination with Drug-eluting Stent
  2. . Drug-coated balloon only
  3. . Drug-eluting stent only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug-coated balloon in combination with drug-eluting stent (Experimental): 40 patients will be treated with a combination of both Pantera® Lux® (Drug Coated Balloon) and Orsiro® (Drug Eluting Stent).
  Interventions: Procedure: Percutaneous Coronary Intervention
- Drug-coated balloon only (Experimental): 40 patients will be treated with Pantera® Lux® (Drug Coated Balloon) only
  Interventions: Procedure: Percutaneous Coronary Intervention
- Drug-eluting stent only (Active Comparator): 40 patients will be treated with a combination of both Pantera® Lux® (Drug Coated Balloon) and Orsiro® (Drug Eluting Stent).
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Percutaneous transluminal coronary angioplasty
  Other Names: PTCA

SUMMARY:
Purpose of this study:

The purpose of the study is to find out whether using a drug coated balloon in combination with a drug-eluting stent is better than the standard practice of using either device on its own. This study is specifically looking at patients with diabetes who have coronary artery disease. This means that their arteries become restricted or blocked, and these restrictions or blockages are called lesions. The study will look at diabetic patients undergoing treatment for lesions in segments of their coronary arteries that have not previously been treated with stents. These are called 'de novo' lesions.

The treatment being investigated:

In this study, we are comparing two devices, either used together or on their own to treat coronary artery disease. These devices are commercially available in Europe and carry the mark. This study is being carried out to compare the effectiveness of combining the two devices or using them individually:

* Pantera® Lux® Paclitaxel Drug Coated Balloon, abbreviated Pantera® Lux® (DCB) A drug coated balloon is a balloon which is covered by an anti-proliferative drug.
* Orsiro® biodegradable polymer Sirolimus Eluting Stent Orsiro® (DES) A stent is a short, wire mesh tube that acts like a scaffold to keep your artery open. A drug eluting stent is coated with medication that reduces the risk of the artery becoming blocked again.

Both drug-eluting stents and drug-coated balloons are used routinely for the treatment of 'de novo' coronary artery disease in Europe.

How will the study be carried out?

This study is being conducted in 4 hospitals across Ireland. We aim to recruit 120 participants s in this study. If you agree to participate in this study and sign the informed consent form, you will be asked to participate in the screening process, which will determine if you meet the conditions to participate in the study.

You will be "randomised" into one of the 3 study groups. Randomisation means that you are put into a group by chance (similarly to the roll of a dice). Neither you nor your doctor can choose the group you will be in. You will not know which group you were placed in until the end of the study. However, your doctor will know which study group you were placed in.

* 40 patients will be treated with Pantera® Lux® (Drug Coated Balloon) only
* 40 patients will be treated with Orsiro® (Drug Eluting Stent) only
* 40 patients will be treated with a combination of both Pantera® Lux® (Drug Coated Balloon) and Orsiro® (Drug Eluting Stent).

If you agree to participate in the study you will be invited to come back for a check-up angiogram 6 months after your procedure to make sure that the treatment has been a success. This is sometimes done in normal clinical practice, but it is not done routinely. You will not be charged for this additional test.

DETAILED DESCRIPTION:
Study Rationale

Stent failure, ISR and TLF remain a significant challenge when considering percutaneous treatment options for de novo CAD in patients with diabetes mellitus. The use of combination treatment with both DCB and DES in this population has not been studied. This study aims to compare the safety and efficacy of a novel combination revascularisation strategy to DCB or DES alone in patients with de novo CAD and diabetes mellitus, a patient group that is at increased risk of TLF compared to patients who do not have diabetes mellitus.

Study Objective

To investigate the efficacy and safety of combination treatment for patients with diabetes mellitus and de novo obstructive CAD undergoing PCI consisting of angioplasty with DCB combined with DES in comparison to single device treatments with either DES or DCB alone, in a randomised, multicentric clinical trial.

Study Design

DUBSTENT-DIABETES is a prospective, randomized, multicentre, assessor-blind, investigator-initiated clinical trial. To investigate the safety and efficacy of combination treatment for patients with de novo CAD undergoing PCI. Consisting of angioplasty with DCB combined with stenting with DES in comparison to single device treatments with either DES or DCB alone.

The study will enrol 120 patients who will be randomized in a 1:1:1 fashion to receive Pantera® Lux® DCB in combination with Orsiro® DES (investigational strategy), or Pantera® Lux® DCB alone, or Orsiro® DES alone (standard of care arm). Subjects will be prospectively enrolled at 4 sites in the Republic of Ireland. In the Pantera® Lux® DCB alone comparator arm, bailout stenting will be allowed under certain criteria. The criteria for bailout stenting will be NHLBI dissection class D to F, and class C at the discretion of the operator. The Freesolveᵀᴹ resorbable magnesium scaffold should be used for bailout stenting to facilitate a leave nothing behind strategy for this comparator arm.

Patients will be screened according to the study inclusion and exclusion criteria (section) prior to coronary angiography. Patients with diabetes mellitus, planned for PCI for de novo obstructive CAD will be eligible. Baseline QCA will be performed to screen patients according to the angiographic inclusion criteria. Subjects who meet all of the study inclusion and exclusion criteria will be eligible for randomisation. Included subjects will then be randomised to either the investigational arm of combination treatment (DCB and DES treatment), or to the comparator arms of DCB treatment, or DES treatment (standard of care arm). Subjects will then receive treatment according to the randomisation.

All procedures will be performed by fully trained operators with several years of interventional experience. All procedures will be performed according to current guidelines and international standards using the Pantera® Lux® DCB and/or the Orsiro® DES. In all patients intravascular imaging is encouraged, but not mandated in the protocol. A pre-specified sub study will take place for 30 subjects who will receive optimal coherence tomography (OCT) imaging.

Baseline characteristics, vital signs, concomitant diseases, cardiovascular risk factors, medication, routine laboratory analyses, ECG data, QCA images and procedural data including periprocedural complications, and follow-up data will be collected.

All included subjects will undergo protocol mandated QCA at 6-months. The primary endpoint of the study, in-segment DS will be assessed by QCA at 6-months follow-up. Key secondary endpoints include TLF, the individual components of TLF (cardiovascular death, non-fatal MI related to the target vessel and unplanned ischaemia-driven TLR). Secondary endpoints will be assessed at 30 days, 6 months and annually up to 5 years. All angiographic endpoints including the primary endpoint will be analysed at Imaging Core Laboratory CVRI Dublin. All clinical events will be adjudicated upon by an independent CEC. The study will be conducted in accordance with the investigation plan, the current version of the Declaration of Helsinki, and national legal and regulatory requirements (2013) (15).

Study Duration

This study will enrol 120 patients in up to 4 investigative centres in the Republic of Ireland over a period of 12 months. Subjects will have follow up QCA performed 6 months after the index QCA. In-person or telephone follow-up appointments will take place at 1 year, then annually up to 5 years after the index procedure. The expected duration of the study is approximately 78 months. This consists of 12 months enrolment followed by 5 years follow up of participants from the time of enrolment of the final participant. An additional 6 months will be permitted for data freeze and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute or chronic coronary syndrome
2. Diagnosis of diabetes
3. Patients undergoing PCI for de novo lesions in native coronary arteries
4. Patients able and willing to provide written informed consent
5. Age ≥ 18 years.
6. Patients able and willing to comply with the study procedures and follow-up.
7. All angiographic inclusion criteria fulfilled:

   1. the lesion has been deemed treatable
   2. the guidewire has crossed the lesion
   3. the lesion has been successfully pre-dilated, where balloon expansion is complete, residual stenosis is less than 50% and thrombolysis in myocardial infarction (TIMI) flow is >2, and there is no evidence of flow-limiting dissection is seen.

Exclusion Criteria:

1. Lesions located at the left main coronary artery.
2. Patient presents with a ST-elevation myocardial infarction (STEMI).
3. Patient with acute cardiac decompensation or acute cardiogenic shock.
4. Patient with impaired renal function (glomerular filtration rate < 30 mL/min/1.73 m2).
5. Severe in-stent calcification that prevents a sufficient expansion of the DCB, unless adequately pre-treated, e.g. with super (high) pressure balloon, rotablation or lithotripsy.
6. Evidence of high-grade dissection (National Heart, Lung, and Blood Institute (NHLBI) class C or greater) at baseline
7. Known hypersensitivity or contraindication to sirolimus, paclitaxel, heparin, aspirin, thienopyridines, or iodinated contrast that cannot be pre-treated.
8. Patients unable to take dual antiplatelet therapy for 6-12 months
9. Pregnant and/or breast-feeding females or females who intend to become pregnant during the time of the study.
10. Subject currently enrolled in other investigational device or drug trial in which the primary endpoint has not yet been reached.
11. Anticipated difficulties to complete the angiographic surveillance.
12. Patient with a life expectancy of less than 12 months.
13. Patients lacking mental capacity (i.e. patients suffering from dementia and others) to provide informed consent.
14. The study will not recruit participants who, in the opinion of the investigator, do not have an adequate understanding of English. Only participants who can fully comprehend the implications of participating in the study will be recruited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2031-08-05 (Estimated)

PRIMARY OUTCOMES:
Percentage Diameter Stenosis | 6 months post PCI (treatment)
  The primary endpoint is percentage diameter stenosis (%DS) of the target lesion segment (target lesion ± 5 mm either side) assessed by QCA at 6 months.

SECONDARY OUTCOMES:
Late Lumen Loss | 6 months
  Late lumen loss assessed by Quantitative Coronary Angiogram (QCA)
Binary Restenosis | 6 months
  Binary Restenosis assessed by Quantitative Coronary Angiogram (QCA)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Byrne, PhD, Study Chair — RCSI University of Medicine and Health Sciences
Locations (1):
- Mater Private Hospital, Dublin, County Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No